CLINICAL TRIAL: NCT06641141
Title: The Feasibility Of Expectant Management Versus Induction At 38 Weeks Among Individuals With Gestational Diabetes Mellitus: A Randomized Controlled Pilot Trial
Brief Title: The Feasibility Of Expectant Management Versus Induction At 38 Weeks Among Individuals With Gestational Diabetes Mellitus: A Randomized Controlled Pilot Trial (EAGER Pilot Trial)
Acronym: EAGER Pilot
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CTO 4937; PJT-191790 (Other Grant/Funding Number: Canadian Institutes of Health Research)
Record Dates: First submitted 2024-10-11; First posted 2024-10-15 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Gestational Diabetes Mellitus (GDM)
Keywords: gestational diabetes mellitus; gestational diabetes; induction; induction of labour
MeSH Terms: conditions — Diabetes, Gestational | interventions — Labor, Induced; Neoadjuvant Therapy

STUDY DESIGN:
Intervention Model Description: This is a multi-centre Prospective Randomized Open-label Blinded Endpoint (PROBE) Pilot Trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Induction of Labour between 38 weeks + 0 days and 38 weeks + 6 days (Experimental): Induction of Labour between 38+0 weeks and 38+6 weeks.
  Interventions: Procedure: Induction of Labour
- Expectant Management (No Intervention): Expectant management without intervention until spontaneous labour, or earlier at the discretion of the attending healthcare provider.

INTERVENTIONS:
Procedure: Induction of Labour — Induction of Labour (IOL) will occur between 38+0 weeks and 38+6 weeks. All participating sites will follow an evidence-based approach for IOL, which may include any of the following: use of prostaglandins, oxytocin, amniotomy, or intracervical balloon catheters with and without extra-amniotic saline infusion for the intervention arm. Participants who are induced in either the intervention or control arms will be managed by their delivery care provider to ensure sufficient time to labour and determine when to proceed to Cesarean delivery. What constitutes a "failed" IOL will be dictated by local clinical practice guidelines and will be informed by the time since IOL (24-48 hours) and/or physician diagnosis of labour dystocia.
  Other Names: IOL; Induction
  Arms: Induction of Labour between 38 weeks + 0 days and 38 weeks + 6 days

SUMMARY:
The EAGER pilot trial is designed to assess the feasibility of a Canadian, multicentre prospective randomized open-label blinded end-point (PROBE) clinical trial addressing whether induction of labour (IOL) at 38 weeks' gestation compared to expectant management (EM) reduces severe perinatal mortality and morbidity among individuals with gestational diabetes mellitus (GDM). Eligible participants will be consented between 32 weeks + 0 days and 38 weeks + 0 days gestation and randomized between 36 weeks + 0 days and 38 weeks + 0 days gestation. Participants will be randomized to one of two arms:

* Intervention Arm: IOL between 38 weeks + 0 days and 38 weeks + 6 days OR
* Control Arm: EM without intervention until spontaneous labour, or earlier if a medical indication arises.

A total of 260 participants (130 per group) will be recruited from Canadian sites, where participants will have 3 study visits:

1. Enrollment and randomization
2. After delivery and up to 72 hours postpartum
3. 6 weeks postpartum At enrollment and randomization, patient-reported baseline and clinical data from medical charts will be collected. Upon admission to hospital for labour and delivery, a blood sample may be collected to assess HbA1C and plasma glucose levels. After delivery and up to 72 hours postpartum, study feasibility will be assessed through patient-reported outcomes and administrative and clinical data. At 6 weeks postpartum, participants will be surveyed for secondary health resource use. Findings from this pilot will inform the design, implementation and feasibility of a future full-scale randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of GDM after 24 weeks of gestation, based on documented 1-step or 2-step screening and diagnostic tests for GDM.
* Singleton fetus at randomization.
* Confirmed live fetus within 24 hours prior to randomization.
* Gestational age between 36 weeks + 0 days and 38 weeks + 0 days inclusive based on an ultrasound in the first or second trimester [≤ 23 weeks + 0 days]. For pregnancies conceived by in vitro fertilization, dating will be based on the embryo age at transfer.
* Cephalic presentation.
* Planning to deliver at a participating site.
* Aged 16 years or older.

Exclusion Criteria:

* Pre-pregnancy diabetes mellitus.
* Any obstetrical/maternal indication for immediate delivery including placenta abruption, abnormal fetal well-being either by non-stress test or biophysical profile, history of venous thromboembolism (VTE) on low molecular weight heparin, pre-existing hypertension, gestational hypertension, preeclampsia, eclampsia, or Hemolysis, elevated liver enzymes and low platelets (HELLP) syndrome at the time of randomization.
* Contraindication to labour and/or vaginal delivery.
* Signs of labour (regular uterine contractions accompanied by cervical dilation and/or effacement) at the time of randomization.
* Significant vaginal bleeding or ruptured membranes at the time of randomization.
* Prior Cesarean delivery.
* Placenta previa, placenta accreta, or vasa previa.
* Cerclage in current pregnancy.
* Known major fetal anomaly (e.g., gastroschisis, congenital heart defects).
* Known oligohydramnios (AFI < 5 or MVP < 2 or no 2 by 2 pocket).
* Known fetal growth restriction (EFW < 3rd percentile).
* Refusal of blood products.
* Use of unregulated substances.

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Participant Recruitment Rate | Within 24 months of randomizing the first participant
  The pilot trial will be considered feasible if least 75% of the target sample can be recruited after 24 months of recruitment. The number of screened, approached, consented and randomized individuals will be recorded to assess feasibility. Recruitment rate will be measured by the proportion of eligible participants enrolled (consented and randomized) into the study.

SECONDARY OUTCOMES:
Appropriateness of eligibility criteria | Within 24 months of randomizing the first participant
  The appropriateness of the eligibility criteria will be assessed. This will be measured as the proportion of screened participants who are excluded overall and per exclusion criterion. It will be reported as numbers (n) and percentages (%).
Participant retention | Within 24 months of randomizing the first participant
  Participant retention will be assessed. This will be measured as the rate of loss to follow-up or withdrawal of consent from randomized participants. It will be reported as numbers (n) and percentages (%).
Non-compliance | Within 24 months of randomizing the first participant
  Participant and healthcare provider non-compliance will be assessed. This will be measured as the proportion of participants who receive off-protocol delivery management, including late IOL. It will be reported as numbers (n) and percentages (%).
Participant satisfaction | Within 24 months of randomizing the first participant
  Participant satisfaction with participating in this study will be assessed. This will be assessed via established surveys: The Labour Agentry Scale, the Study Participant Feedback Questionnaire and the Decisional Regret Scale.
Suitability of maternal and neonatal clinical endpoints. | Within 24 months of randomizing the first participant
  Suitability of maternal and neonatal clinical endpoints for an eventual full-scale trial will be assessed. This will be assessed based on expert consultation (clinical experts and individuals with lived experience) and will account for the rate of occurrence of severe maternal and neonatal outcomes, and quality and completeness of collected data.

CONTACTS AND LOCATIONS:
Overall Officials: Mark C Walker, MD, MSc, MHM, Principal Investigator — Ottawa Hospital Research Institute; Darine El-Chaâr, MD, FRCS(C), MSc, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada